CLINICAL TRIAL: NCT01043692
Title: Acceptability of a Strategy Including Acupuncture in the Treatment of MusculoSkeletal Pain in Hospitalised Elderly
Brief Title: Acceptability of an Acupuncture Intervention in Painful Elderly
Acronym: ACUPUNCTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-AOO534-47
Record Dates: First submitted 2009-12-21; First posted 2010-01-07 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2009-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain > 3 months; Acupuncture; Acceptability; Geriatrics
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Acupuncture in the Treatment of MUSCULOSKELETAR Pain in Hospitalised Elderly
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture in the Treatment of MUSCULOSKELETAR Pain in Hospitalised Elderly

SUMMARY:
The aim is to investigate the feasibility and efficacy of an acupuncture intervention on persistent MusculoSkeletar pain in a long-term geriatric hospital care ward population. The main issue is the acceptability of this type of complementary and alternative medicine in older people, although the efficacy on pain is assessed too.

DETAILED DESCRIPTION:
The first 60 patients wanting to participate are enrolled. For the impaired patients, family or legal representing is solicited. The Regional Ethic Committee agreement was granted. The intervention consists in 8 acupuncture sessions.

Evaluation

* Acceptability : the proportion of patients who complete the whole treatment ; the acceptability at each acupuncture session is recorded.
* Pain : Dolorous Scale . The evaluation is based on pre and post treatment variations. As a high proportion of patients have cognitive impairment, the behavioural pain scale "dolorous" has been chosen after staffs training for all patients, although "extra " auto evaluation is used when possible (EVS). Evaluation takes place after 5 sessions and after the end of the intervention as well as 2 and 4 weeks after the interventionProfessional carers' satisfaction is recorded.

ELIGIBILITY:
Inclusion Criteria:

* age > 60 years
* chronic musculoskeletal pain
* follow up 10 weeks
* patient or legal representative's agreement to participate and to the informatics treatment of the data

Exclusion Criteria:

* acute pain
* exclusive neurological pain
* coagulation disorders or anticoagulant curative treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Taux acceptability of the totality of treatment | 6 months

SECONDARY OUTCOMES:
Participation rate | every visit
Motives behind the acceptance or rejection | at Visit 0 to 8
Pain decrease assessment : DOLOPLUS score (observer-assessed evaluation of pain) before/ater intervention, for all the patients Simple descriptive pain intensity scale (VS) (self assessment evaluation of pain) for communicative patients | at Visit 0, 6, 9, 10 and 11
Pain therapeutic's decrease | every visit
Patient's benefit - Carers satisfaction (questionnaire) | at Visit 0,6, 9, 10 and 11

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France COUILLIOT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- HOPITAL RENE MURET BIGOTTINI - Dpt Interhosp. Santé Pub., Sevran, France

REFERENCES:
- [Result] Couilliot MF, Darees V, Delahaye G, Ercolano P, Carcaille M, Vytopilova P, Tenenbaum B, Vicaut E. Acceptability of an acupuncture intervention for geriatric chronic pain: an open pilot study. J Integr Med. 2013 Jan;11(1):26-31. doi: 10.3736/jintegrmed2013005. PMID 23464643